CLINICAL TRIAL: NCT00765219
Title: Treating Late-life GAD in Primary Care: Enhancing Outcomes and Translational Value
Brief Title: Cognitive Behavior Treatment of Older Adults With Generalized Anxiety Disorder in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Melinda Stanley, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H23798; R01MH053932-10A1 (NIH)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Geriatric
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): CBT with ACS
  Interventions: Behavioral: CBT
- 2 (Experimental): CBT with Counselor
  Interventions: Behavioral: CBT
- 3 (Active Comparator): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: CBT — 10-12 weekly sessions of CBT in person or over the telephone.
  Other Names: Cognitive Behavior Treatment, Cognitive Behavior Therapy
  Arms: 1; 2
Other: Usual Care — Treatment as usual provided by participants' physician(s)
  Other Names: Treatment as Usual
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether cognitive behavior treatment (CBT) can be delivered effectively by providers of different expertise levels in adults age 60 and older in a primary care setting.

DETAILED DESCRIPTION:
Generalized Anxiety Disorder (GAD) is one of the most common anxiety disorders among older adults. Anxiety in older adults is associated with decreased physical activity, poorer self-perceptions of health, decreased life satisfaction, and increased loneliness. Because many older adults with anxiety seek assistance in a medical setting, treatment has been primarily pharmacological. There is, however, limited evidence of the effectiveness of psychotropic medications in later life. Given the potential difficulties in prescribing psychotropic medications in later life(e.g., increased adverse effects, potential drug interactions), psychosocial treatments may be important alternatives or adjuncts.

The treatment phase of this study lasts 6 months, during which patients will be randomly assigned to either cognitive behavior treatment (CBT) with an Anxiety Clinic Specialist (ACS) or Counselor or to Usual Care (UC). All participants will complete telephone assessments at baseline, 1, 2, and 3 months during the treatment phase. During the first 12 weeks, those assigned to CBT will also complete 10-12 weekly sessions, either in person or over the telephone. During the second 12 weeks, CBT patients will receive follow-up telephone booster calls, weekly for the first 4 weeks and biweekly for the last 8 weeks. During the treatment phase, UC participants will receive no treatment from study clinicians but will continue to receive their usual care from their current medical providers.

At 6 months, all participants will complete a telephone assessment. CBT patients will enter a one year follow-up period, with telephone assessments at 12 and 18 months. UC participants will be offered the option to receive brief CBT after completion of the 6 month telephone assessment. Those who choose to participate in CBT will complete telephone assessments at 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older
* Principal or Co-principal GAD diagnosis
* Patient at participating clinic

Exclusion Criteria:

* Active suicidal intent
* Current psychosis or bipolar disorder
* Substance abuse within the past month
* Cognitive impairment according to a Mini Cog screener score of 3 or lower

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2008-05; Primary Completion 2013-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Anxiety | 18 months

SECONDARY OUTCOMES:
Depression | 18 months
Sleep quality | 18 months
Use of alcohol | 18 months
Functional and health status | 18 months
Quality of life | 18 months
Pain | 18 months
Satisfaction with CBT and general health care | 18 months
Service utilization | 18 months
Use of psychotropic medications | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Melinda A. Stanley, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Center for Quality of Care and Utilization Studies, Houston, Texas, United States

REFERENCES:
- [Derived] Freshour JS, Amspoker AB, Yi M, Kunik ME, Wilson N, Kraus-Schuman C, Cully JA, Teng E, Williams S, Masozera N, Horsfield M, Stanley M. Cognitive behavior therapy for late-life generalized anxiety disorder delivered by lay and expert providers has lasting benefits. Int J Geriatr Psychiatry. 2016 Nov;31(11):1225-1232. doi: 10.1002/gps.4431. Epub 2016 Feb 28. PMID 26923925
- [Derived] Barrera TL, Cully JA, Amspoker AB, Wilson NL, Kraus-Schuman C, Wagener PD, Calleo JS, Teng EJ, Rhoades HM, Masozera N, Kunik ME, Stanley MA. Cognitive-behavioral therapy for late-life anxiety: Similarities and differences between Veteran and community participants. J Anxiety Disord. 2015 Jun;33:72-80. doi: 10.1016/j.janxdis.2015.04.005. Epub 2015 May 7. PMID 26005839